CLINICAL TRIAL: NCT04566783
Title: Identification of Etiopathological and Clinical Factors in Persistent Genital Arousal Disorder: The iPGAD-Study
Brief Title: Identification of Etiopathological and Clinical Factors in Persistent Genital Arousal Disorder
Acronym: iPGAD
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 8589_BO_S_2019
Record Dates: First submitted 2020-06-09; First posted 2020-09-28 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Restless Genital Syndrome; Sexual Arousal Disorder; Orgasmic Disorder; Psychosexual Disorder
Keywords: Persistant Genital Arousal Disorder; PGAD
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Neurologic Examination; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women and men fulfilling PGAD-criteria: Inclusion criteria:
  - Female and male patients or subjects between 18-65 years of age fulfilling the diagnostic criteria of persistent genital arousal disorder (PGAD) according to Leiblum & Nathan (2001).
  Exclusion criteria:
  - Any exclusion criteria for magnetic resonance imaging (MRI), mental retardation, severe and acute somatic or mental disease such as acute psychosis, brain damage, Alzheimer's disease, severe bacterial infection requiring immediate medical treatment.
  Age:
  - 18 - 65 years of age
  Gender:
  - Female and male subjects
  Interventions: Diagnostic Test: Psychological/psychiatric examination; Diagnostic Test: Neurological examination; Diagnostic Test: Gynecological/urological examination; Diagnostic Test: Laboratory assessment; Diagnostic Test: Structural and Functional Magnetic Resonance Imaging
- Controls: Inclusion criteria:
  - Age and education matched healthy controls.
  Interventions: Diagnostic Test: Psychological/psychiatric examination; Diagnostic Test: Neurological examination; Diagnostic Test: Gynecological/urological examination; Diagnostic Test: Laboratory assessment; Diagnostic Test: Structural and Functional Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Psychological/psychiatric examination — Thorough diagnostic and (neuro)psychological assessment using standardized clinical interviews (e.g. MINI, SOMS) as well as questionnaires assessing sexual function (e.g. SIS/SES), depression and anxiety (HADS), childhood trauma (CTQ) and life quality (WHOQOL-BREF). In a semi-structured interview sociodemographic data, drug history and sexual characteristics are captured.
Diagnostic Test: Neurological examination — Standardized clinical neurological examination as well as neurophysiological measurements (Pudenus-SEP, ENoG, clinical EEG).
Diagnostic Test: Gynecological/urological examination — Standard clinical investigation including ultrasound of the genital organs will be conducted to look for any somatic pathology (e.g. varices, tumors).
Diagnostic Test: Laboratory assessment — Blood sample will be analyzed to evaluate (epi-)genetic markers of increased central excitability or decreased inhibition including specific parameters of the serotonin-, dopamine- and endocannabinoid system.
Diagnostic Test: Structural and Functional Magnetic Resonance Imaging — 1. Structural MRI of the pelvis is conducted to rule out any anatomical pathologies underlying PGAD (e.g. varices).
  2. Structural MRI of the lumbosacral spinal cord to look for any pathologies on the spinal level, especially spinal level S2-4 (e.g. Tarlov cysts).
  3. High-resolution structural MRI (T1) including brain stem will be applied to all participants in order to explore alterations in gray matter volume or density.
  4. Structural differences in white matter will be assessed using a high-resolution DTI sequence. In addition to standard voxel-wise comparison of DTI derived parameters for white matter microstructural integrity, a tractography-based analysis will test for alterations in structural connectivity.
  5. Resting-state functional MRI including brain stem scans will evaluate abnormal brain circuitry at rest (resting-state functional connectivity, RSFC).
  6. Functional MRI to assess brain response towards sexual cue reactivity.

SUMMARY:
Investigation of (possible etiological) factors associated with PGAD symptomatology as well as description of comorbid disorders subjects with PGAD.

Persistent genital arousal disorder (PGAD) is a presumably rare, although debilitating condition, which was first defined at the beginning of this century and has not yet found consideration by any of the international classification systems of diseases. PGAD is commonly characterized by persistent and unwanted sensations of genital arousal which are not related to subjective feelings of sexual desire or arousal. Affected patients which are predominantly women can suffer tremendously. The lack of basic research on the etiology of PGAD leads to insufficient therapeutical approaches.

DETAILED DESCRIPTION:
The entire approach is of multimodal and explorative nature as only very limited information on this disease is available so far (hypotheses generating). Moreover, the aim of the study is to characterize PGAD patients in terms of their biography (e.g. trauma), comorbidities and life quality.

Clinical assessment:

* Psychological/psychiatric examination
* Neurological examination
* Gynecological/urological examination
* Laboratory assessment
* Structural and Functional Magnetic Resonance Imaging

General Hypotheses:

1. There is a morphological correlate of PGAD that affects or represents a neuronal structure leading to altered perception of genital sensation (e.g. Tarlov cysts, varices, …).
2. There is a functional correlate of PGAD in the central nervous system (CNS) indicating a hyperfunction (excitation or disinhibition) or hypofunction (inhibition) of specific brain areas including hypothalamus, sensory cortex of the genitals and secondary brain areas, brain stem centers (e.g. raphe nuclei) and others.
3. Patients with PGAD show an elevated rate of previous pharmacological treatment with drugs that may alter the central processing of sexual/genital perception or reveal a specific pattern of comorbid diseases (e.g. affective or somatoform disorders) that may predispose other disorders such as PGAD, pain disorders etc.

Expected results and exploitation:

The proposed project will help to identify clinical and neurobiological correlates of persistent genital arousal (PGAD) and will provide

1. a deeper clinical, (neuro)psychological and (neuro)biological understanding of PGAD
2. help to identify related etiopathological mechanisms of PGAD
3. inform clinicians and (sex) therapists on diagnostic issues and promising treatment targets in PGAD derived from comprehensive clinical and experimental measures
4. stimulate further neurobiological and clinical research in the field of PGAD, leading to further national and international cooperation and applications
5. a considerable number of publications in leading scientific journals and raise awareness of a rare disease not only among all clinicians dealing with sexual problems but also general practitioners and others.

Objective(s):

Investigation of (possible etiological) factors associated with PGAD symptomatology as well as description of comorbid disorders subjects with PGAD.

Statistical Analysis:

Clinical (psychological, neurological and gynecological/urological) data is analyzed using a descriptive approach of frequencies and mean values of diverse clinical findings as well as a group comparison (patients versus healthy controls) using respective statistical analyses such as ttests, chi-square test and others after having tested for normal distribution where necessary. MRT data is analyzed using state-of-the-art special software (SPM) including group comparisons.

Sample Size Justification:

This is a cross-sectional study of a rare disease. At MHH usually 10 new patients occur per year. The investigator tries to include as many patients as possible and will probably achieve higher numbers by advertising the study and using data banks of already existing cases. Due to the presumably rare number of people affected with PGAD and the very few existing publications which are mostly case reports and the even fewer PGAD related MRI data a statistically neat sample size computing is not simple. The investigator cannot refer to prior carried out PGAD related MRI studies and to publications mentioning PGAD sample sizes. However, for MRI studies methodological work investigating the reliability of statistical effect in fMRI studies exist. An article by Thirion in 2007 shows that a sample size between 20 and 30 subjects per group is sufficient to detect statistical effects. This is also in accordance with common practice in fMRI aiming at at least 20 subject per group at which results become quite stable (Murphy & Garavan 2004) Thus, the investigator aims at a sample size of 25 subjects per group. To account for potential dropouts (~10%, mainly due to excessive head movement in the MRI scanner) it is planned to include approximately 30 subjects per group.

Discussion of Perceived / Expected Risks and Benefits:

When considering all exclusion criteria for MRI there are no risks known for using a magnetic resonance imaging system. Clinical and (neuro)psychological testing might be perceived stressful by some participants and therefore may lead to a temporary increase in blood pressure and/or heart rate that will normally end after testing. Clinical examination (neurological and gynecological/urological) might lead to discomfort in some participants. Besides the neurological examination which can result in uncomfortable feelings (e.g. minor pain) during the ENoG-testing and Pudendus-SEP and that will normally end immediately after testing the clinical examination is pain-free. Blood Sampling might be painful and lead to hematoma. The amount of blood is low (approx. 30ml). Any serious damage to the organism during clinical examination and blood sampling is very unlikely.

ELIGIBILITY:
Inclusion Criteria:

* female and male subjects
* must be between 18-65 years of age
* must fulfill the diagnostic criteria of persistent genital arousal disorder (PGAD) according to Leiblum & Nathan (2001)
* controls must be healthy and matched in accordance with age and education.

Exclusion Criteria:

* any exclusion criteria for magnetic resonance imaging
* mental retardation
* severe somatic or mental disease such as acute psychosis, brain damage, Alzheimer disease
* severe bacterial infection requiring immediate medical treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * female and male patients or subjects between 18-65 years of age fulfilling the diagnostic criteria of persistent genital arousal disorder (PGAD) according to Leiblum & Nathan (2001).
  * additionally, age and education matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
General outcome and target: Identification of clinical and neurobiological correlates of persistent genital arousal (PGAD) | Data collection and avaluation through study completion. Data collection (examinations) will take 1 day (max 2) per subject. Data evaluation of all collected data will take about 1 year. Publication of findings will be an ongoing process afterwards.
  1. gather a deeper clinical, (neuro)psychological and (neuro)biological understanding of PGAD
  2. help to identify related etiopathological mechanisms of PGAD
  3. inform clinicians and (sex) therapists on diagnostic issues and promising treatment targets in PGAD derived from comprehensive clinical and experimental measures
  4. stimulate further neurobiological and clinical research in the field of PGAD, leading to further national and international cooperation and applications
  5. publish a considerable number of publications in leading scientific journals and raise awareness of a rare disease not only among all clinicians dealing with sexual problems but also general practioners and others.
Questionnaires: Psychological/Psychiatric, neurological and gynecological/urological assessments | Data collection and avaluation through study completion. Data collection (examinations) will take 1 day (max 2) per subject. Data evaluation of all collected data will take about 1 year.
  Assessing sexual function (e.g. SIS/SES), depression and anxiety (HADS), childhood trauma (CTQ) and life quality (WHOQOL-BREF). In a semi-structured interview sociodemographic data, drug history and sexual characteristics are captured.
Clinical examinations: Psychological/Psychiatric, neurological and gynecological/urological assessments | Data collection and avaluation through study completion. Data collection (examinations) will take 1 day (max 2) per subject. Data evaluation of all collected data will take about 1 year.
  1. Neuro)psychological assessment using standardized clinical interviews (e.g. MINI, SOMS).
  2. Neurological examination: Standardized clinical neurological examination as well as neurophysiological measurements will be conducted (Pudenus-SEP, ENoG, clinical EEG).
  3. Gynecological/urological examination: Standard clinical investigation including ultrasound of the genital organs will be conducted to look for any somatic pathology (e.g. varices, tumors).
Clinical and experimental imaging (MRI, fMRI) | Data collection and avaluation through study completion. Data collection (examinations) will take 1 day (max 2) per subject. Data evaluation of all collected data will take about 1 year.
  1. Structural MRI of the pelvis is conducted to rule out any anatomical pathologies underlying PGAD (e.g. varices).
  2. Structural MRI of the lumbosacral spinal cord to look for any pathologies on the spinal level (esp. spinal level S2-4 (e.g. Tarlov cysts)).
  3. High-resolution structural MRI (T1) including brain stem will be applied to all participants in order to explore alterations in gray matter volume or density.
  4. Structural differences in white matter will be assessed using a high-resolution DTI sequence. In addition to standard voxel-wise comparison of DTI derived parameters for white matter microstructural integrity, a tractography-based analysis will test for alterations in structural connectivity.
  5. Resting-state functional MRI including brain stem scans will evaluate abnormal brain circuitry at rest (resting-state functional connectivity, RSFC).
  6. Functional MRI to assess brain response towards sexual cue reactivity.
Laboratory assessments (blood samples) | Data collection and avaluation through study completion. Data collection (examinations) will take 1 day (max 2) per subject. Data evaluation of all collected data will take about 1 year.
  Blood sample will be analyzed to evaluate (epi-)genetic markers of increased central excitability or decreased inhibition including specific parameters of the serotonin-, dopamine- and endocannabinoid system

CONTACTS AND LOCATIONS:
Overall Officials: Tillmann Prof. Krüger, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leiblum SR, Nathan SG. Persistent sexual arousal syndrome: a newly discovered pattern of female sexuality. J Sex Marital Ther. 2001 Jul-Sep;27(4):365-80. doi: 10.1080/009262301317081115. PMID 11441520